CLINICAL TRIAL: NCT03567174
Title: Building on Needle Exchange to Optimize Prevention & Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Baltimore City Health Department (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00147873; R01DA045556 (NIH)
Record Dates: First submitted 2018-06-12; First posted 2018-06-25 (Actual); Results first posted 2022-12-27 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Intravenous Drug Usage; HIV/AIDS
Keywords: hepatitis C
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hepatitis C

STUDY DESIGN:
Intervention Model Description: Cluster-randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated care van (ICV) (Experimental): ICV visits neighborhoods served by the mobile syringe service program weekly. ICV provides a range of services targeted to people who inject drugs - HIV testing, HCV testing, PrEP, MAT, wound care, case work services, on-site medical management and linkage.
  Interventions: Other: Integrated care van (ICV)
- Control (No Intervention): No additional services provided.

INTERVENTIONS:
Other: Integrated care van (ICV) — Structural service delivery intervention
  Arms: Integrated care van (ICV)

SUMMARY:
There are several biomedical interventions that can help people who inject drugs (particularly those with or at risk for HIV), but these services often do not get to the people most in need. In this project investigators propose to determine if delivery of these services to PWID by an integrated care van that is linked to a mobile syringe service program improves clinical outcomes, is feasible and sustainable, and is cost-effective.

DETAILED DESCRIPTION:
Biomedical interventions that have direct applicability to people who inject drugs (PWID) have flourished over the past 15 years (HIV treatment as prevention, pre-exposure prophylaxis, office-based medication-assisted treatment (MAT) with buprenorphine, and hepatitis C virus (HCV) treatment with direct acting agents). However, penetration of these interventions among PWID is low relative to the potential benefits. Syringe service programs (SSP) are an essential risk reduction service for PWID, and represent the outermost reach of public health services for this population. The Baltimore City Health Department (BCHD) and investigators at Johns Hopkins University are developing a dedicated integrated care van (ICV) to complement the city's mobile SSP, with the goals of optimizing the HIV care cascade in HIV-positive clients and extending needed biomedical interventions to PWID. A nurse practitioner, case worker, and peer navigators will engage HIV-positive clients (known and newly diagnosed) and collaborate closely with local HIV clinics to promote progress toward durable viral suppression. To support the ICV's role in HIV care facilitation, investigators propose an innovative application of the Center for Disease Control (CDC)-sponsored "Data to Care" initiative - a multi-source health service database designed to assist health departments track the HIV care cascade in real time. Additionally, the ICV will provide rapid HIV testing, PrEP screening and initiation, buprenorphine-based MAT, HCV testing and referrals to treatment, and wound care. Using a cluster-randomized trial design, investigators propose to determine whether the ICV intervention advances the HIV care cascade among HIV-positive PWID, improves the Pre-Exposure Prophylaxis (PrEP) continuum, and increases uptake of MAT and HCV treatment (Aim 1). Additionally, investigators will examine the implementation of the ICV intervention using a mixed methods approach among PWID, local/state public health stakeholders, and medical providers to examine the intervention's feasibility, acceptability, coverage, fidelity, and sustainability (Aim 2). Finally, investigators will determine the incremental cost-effectiveness of the ICV intervention (Aim 3). Investigators have assembled a multi-disciplinary team with methodological expertise in PWID interventions and cost-effectiveness evaluations, and longstanding collaboration with investigators' partners at the BCHD.

ELIGIBILITY:
Inclusion Criteria:

* If HIV-positive: report history of injection drug use
* If HIV-negative: injected drugs ≥ 4 days in the last 30 days or shared a needle or syringe in the last 6 months

Exclusion Criteria:

* Not competent to provide written informed consent
* Not willing or able to provide a blood specimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2022-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory M Lucas, MD, Principal Investigator — Johns Hopkins University; Kathleen Page, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Baltimore City Syringe Service Program Neighborhood sites, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Willing to share de-identified Individual Participant Data (IPD) with researchers that approach our team with an acceptable proposal.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 19 syringe service program (SSP) sites from Baltimore City Health Department were considered for the trial. The 13 sites with the largest numbers of clients in 2017 were initially selected, and one of those 13 was eliminated because it already offered some services planned for the intervention. The remaining 12 sites were paired based on client demographics, SSP client non-overlap between sites, and SSP staff opinions about the similarities of sites.
Units Other Than Participants: Study Sites
Groups:
- Integrated Care Van (ICV): ICV visits neighborhoods served by the mobile syringe service program weekly. ICV provides a range of services targeted to people who inject drugs - HIV testing, hepatitis C virus (HCV) testing, Pre-Exposure Prophylaxis (PrEP), Medication-Assisted Treatment (MAT), wound care, case work services, on-site medical management and linkage.
  Integrated care van (ICV): Structural service delivery intervention
Period: Overall Study
Arm/Group | Integrated Care Van (ICV) | Control
Started | 360; 6 Study Sites | 360; 6 Study Sites
V7 Follow-up | 268; 6 Study Sites | 243; 6 Study Sites
V14 Follow-up (Pre-COVID) | 79; 2 Study Sites | 70; 2 Study Sites
COVID Phone Surveys | 164; 6 Study Sites | 155; 6 Study Sites
V14 Follow-up (Post-COVID) | 92; 4 Study Sites | 85; 4 Study Sites
Completed | 171; 6 Study Sites | 155; 6 Study Sites
Not Completed | 189; 0 Study Sites | 205; 0 Study Sites
Not completed — Death | 24 | 31
Not completed — Lost to Follow-up | 165 | 174

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Integrated Care Van (ICV) | Control | Total
Number analyzed (Participants) | 360 | 360 | 720
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 51.5 [41 to 57] | 48 [38 to 54] | 50 [39 to 55]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 226 | 218 | 444
  Female | 134 | 142 | 276
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 10 | 17
  Not Hispanic or Latino | 352 | 350 | 702
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 4 | 8
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 270 | 253 | 523
  White | 75 | 88 | 163
  More than one race | 8 | 11 | 19
  Unknown or Not Reported | 0 | 1 | 1
Composite PWID Score (Service Access, Risk Behaviors, Adverse Outcomes) [Mean (Standard Deviation); unit: units on a scale] — We developed a scoring rubric based on World Health Organization (WHO) guidelines for evidence-based PWID services, a predictive risk model for HIV seroconversion among PWID developed by the Baltimore-based ALIVE study, the HCV care continuum, and the overdose epidemic. In the score, points are allocated on the basis of failure to access evidence-based services, riskier behaviors, and adverse outcomes.
  The score is based on self-report, biomarker testing, and medical record review, and ranges from 0 to 15, with higher scores indicating worse overall status.
  units on a scale | 7.32 (1.75) | 7.37 (1.94) | 7.35 (1.85)

OUTCOME MEASURES:

1. Primary Outcome: Composite PWID Score (Service Access, Risk Behaviors, Adverse Outcomes)
Description: To capture the multifaceted nature of the ICV intervention and the array of health issues relevant to PWID, we developed a scoring rubric based on World Health Organization (WHO) guidelines for evidence-based PWID services, a predictive risk model for HIV seroconversion among PWID developed by the Baltimore-based ALIVE study, the HCV care continuum, and the overdose epidemic. In the scoring rubric, points are allocated on the basis of failure to access evidence-based services, riskier behaviors, and adverse outcomes.
  This outcome will be assessed in all participants at all time points. The score is based on self-report, biomarker testing, and medical record review, and ranges from 0 to 15, with higher scores indicating worse overall status.
Time Frame: Between baseline visit and the V7 follow-up visit at 7 months
Population: Subset of participants who had calculated composite outcome scores at the V7 visit: participants who either completed the V7 follow-up visit or died before completing the V7 follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Integrated Care Van (ICV) | Control
Number analyzed (Participants) | 272 | 250
units on a scale | 5.34 (2.35) | 5.64 (2.56)
Statistical Analysis 1: Comparison: Integrated Care Van (ICV) vs Control; Test type: Superiority; p = 0.125, Mixed Models Analysis; Mean Difference (Net) = -0.306, 95% CI 2-sided [-0.697 to 0.085]

2. Secondary Outcome: HIV Care Continuum
Description: This outcome will be assessed in HIV-positive participants at all time points. The score is based on self-report and biomarker testing, and ranges from 0 to 2 with higher scores indicating poorer HIV care engagement.
  Participants with viral load suppression (HIV RNA <20 c/mL) are counted and assigned a score=0; those with non-suppressed viral load but who took antiretroviral drugs in the prior 30 days or who had a visit with an HIV care provider in the prior 6 months are counted and assigned a score=1; those with non-suppressed viral load, and who did not take antiretroviral drugs (ARVs) in the prior 30 days and did not have a visit with an HIV care provider in the prior 6 months are counted and assigned a score=2. The counts of participants will be reported for this outcome measure and the associated score will be factored into the primary composite outcome.
Time Frame: Between 6 months prior to and the V7 follow-up visit at 7 months
Population: Subset includes HIV-positive participants who completed the V7 follow-up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Integrated Care Van (ICV) | Control
Number analyzed (Participants) | 32 | 33
Participants
  Suppressed (HIV RNA undetectable) | 13 | 19
  Not suppressed, ARVs in prior 30 days or provider visit last 6 months | 18 | 10
  Not suppressed, no ARVs and no provider visit last 6 months | 1 | 4

3. Secondary Outcome: HIV Testing
Description: This outcome will be assessed in HIV-negative participants at all time points. The score is based on self-report and biomarker testing, and ranges from 0 to 1 with higher scores indicating poorer HIV care engagement.
  Participants who had an HIV test in the prior 6 months will be counted and assigned a score=0; those who did not have an HIV test in the prior 6 months will be counted and assigned a score=1. The counts of participants will be reported for this outcome measure and the associated score will be factored into the primary composite outcome.
Time Frame: Between 6 months prior to and the V7 follow-up visit at 7 months
Population: Subset of participants who were HIV-negative at both baseline and V7 follow-up visits and completed the V7 follow-up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Integrated Care Van (ICV) | Control
Number analyzed (Participants) | 236 | 210
Participants
  Had an HIV test in the prior 6 months | 234 | 202
  Did not have an HIV test in the prior 6 months | 2 | 8

4. Secondary Outcome: Pre-exposure Prophylaxis (PrEP) Continuum
Description: This outcome will be assessed in HIV-negative participants at all time points. The score is based on self-report, and ranges from 0 to 1 with higher scores indicating poorer engagement with PrEP.
  Participants who used PrEP in the prior 6 months are counted and assigned a score=0; those who did not use PrEP in the prior 6 months are counted and assigned a score=1. The counts of participants will be reported for this outcome measure and the associated score will be factored into the primary composite outcome.
Time Frame: Between 6 months prior to and the V7 follow-up visit at 7 months
Population: Subset of participants who were HIV-negative and completed the V7 follow-up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Integrated Care Van (ICV) | Control
Number analyzed (Participants) | 236 | 210
Participants
  Used PrEP in the prior 6 months | 0 | 4
  Did not use PrEP in the prior 6 months | 236 | 206

5. Secondary Outcome: HCV Care Continuum
Description: This outcome will be assessed in HCV-positive participants at all time points. The score is based on self-report and biomarker testing, and ranges from 0 to 2 with higher scores indicating poorer engagement with HCV care.
  Participants successfully treated for HCV with undetectable HCV RNA are counted and assigned a score=0; those who have detectable HCV RNA but who have been evaluated or treated for HCV in the prior 6 months are counted and assigned a score=1; those who have detectable HCV RNA, have not been treated or evaluated in the prior 6 months are counted and assigned a score=2. The counts of participants will be reported for this outcome measure and the associated score will be factored into the primary composite outcome.
Time Frame: Between 6 months prior to and the V7 follow-up visit at 7 months
Population: Subset includes HCV-positive participants (including viremic or non-viremic with treatment completion) who completed the V7 follow-up visit
Measure: Count of Participants; unit: Participants
Arm/Group | Integrated Care Van (ICV) | Control
Number analyzed (Participants) | 145 | 103
Participants
  Successfully treated for HCV with undetectable HCV RNA | 34 | 20
  Detectable HCV RNA but who have been evaluated or treated for HCV in the prior 6 months | 36 | 25
  Detectable HCV RNA, have not been treated or evaluated in the prior 6 months | 75 | 58

6. Secondary Outcome: HCV Testing
Description: This outcome will be assessed in HCV-negative participants and HCV-antibody positive participants who spontaneously cleared the infection without completing treatment at all time points. The score is based on self-report and biomarker testing, and ranges from 0 to 1 with higher scores indicating poorer HIV care engagement.
  Participants who had an HCV test in the prior 6 months are counted and assigned a score=0; those who did not have an HCV test in the prior 6 months are counted and assigned a score=1. The counts of participants will be reported for this outcome measure and the associated score will be factored into the primary composite outcome.
Time Frame: Between 6 months prior to and the V7 follow-up visit at 7 months
Population: Subset includes HCV-antibody negative participants and HCV-antibody positive participants who spontaneously cleared the infection without completing treatment and completed the V7 follow-up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Integrated Care Van (ICV) | Control
Number analyzed (Participants) | 122 | 139
Participants
  Had an HCV test in the prior 6 months | 65 | 66
  Did not have an HCV test in the prior 6 months | 57 | 73

7. Secondary Outcome: Medication for Opioid Use Disorder (MOUD) Use
Description: This outcome will be assessed in all participants at all time points. The score is based on self-report, and ranges from 0 to 1.
  Participants who used MOUD in the prior 6 months are counted and assigned a score=0; those who have not used MOUD in the prior 6 months are counted and assigned a score=1. The counts of participants will be reported for this outcome measure and the associated score will be factored into the primary composite outcome.
Time Frame: Between 6 months prior to and the V7 follow-up visit at 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Integrated Care Van (ICV) | Control
Number analyzed (Participants) | 268 | 243
Participants
  Used MOUD in the prior 6 months | 165 | 134
  Have not used MOUD in the prior 6 months | 103 | 109

8. Secondary Outcome: Syringe Service Program (SSP) Use
Description: This outcome will be assessed in participants who report injection drug use in the prior 6 months, at all time points. The score is based on self-report, and ranges from 0 to 1 with higher scores indicating poorer engagement in risk reduction services.
  Participants who used an SSP in the prior 6 months are counted and assigned a score=0; those who did not use an SSP in the prior 6 months are counted and assigned a score=1. The counts of participants will be reported for this outcome measure and the associated score will be factored into the primary composite outcome.
Time Frame: Between 6 months prior to and the V7 follow-up visit at 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Integrated Care Van (ICV) | Control
Number analyzed (Participants) | 268 | 243
Participants
  Used an SSP in the prior 6 months | 223 | 208
  Did not use an SSP in the prior 6 months | 45 | 35

9. Secondary Outcome: Naloxone Overdose Kit
Description: This outcome will be assessed in all participants at all time points. The score is based on self-report, and ranges from 0 to 1 with higher scores indicating poorer engagement in risk reduction services.
  Participants who possess a naloxone overdose kit that is usually accessible when they use drugs (i.e, where they usually use drugs) are counted and assigned a score=0; those who do not possess a naloxone overdose kit that is in an accessible location are counted and assigned score=1. The counts of participants will be reported for this outcome measure and the associated score will be factored into the primary composite outcome.
Time Frame: Between 6 months prior to and the V7 follow-up visit at 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Integrated Care Van (ICV) | Control
Number analyzed (Participants) | 268 | 243
Participants
  Possess a naloxone overdose kit that is in an accessible location (where they usually use drugs) | 164 | 157
  Do not possess a naloxone overdose kit that is usually accessible when they use drugs | 104 | 86

10. Secondary Outcome: Injection Drug Use
Description: This outcome will be assessed in all participants at all time points. The score is based on self-report and ranges from 0 to 1 with higher scores indicating riskier behavior.
  Participants who did not inject drugs in the prior 6 months are counted and assigned a score=0; those who did inject drugs in the prior 6 months are counted and assigned a score=1. The counts of participants will be reported for this outcome measure and the associated score will be factored into the primary composite outcome.
Time Frame: Between 6 months prior to and the V7 follow-up visit at 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Integrated Care Van (ICV) | Control
Number analyzed (Participants) | 268 | 243
Participants
  Did not inject drugs in the prior 6 months | 108 | 85
  Did inject drugs in the prior 6 months | 160 | 158

11. Secondary Outcome: Recent Drug Use
Description: This outcome will be assessed in all participants at all time points. The score is based on biomarker testing and ranges from 0 to 1 with higher scores indicating riskier behavior.
  Participants who have a negative urine drug test for selected drugs are counted and assigned a score=0; those who have a positive urine drug test for selected drugs are counted and assigned a score=1. The counts of participants will be reported for this outcome measure and the associated score will be factored into the primary composite outcome.
  Selected drugs include the primary drug or metabolites of fentanyl, heroin, cocaine, or amphetamines.
Time Frame: Between 6 months prior to and the V7 follow-up visit at 7 months
Population: Subset of participants who completed a V7 follow-up visit and had available urine toxicology result. Two participants did not have urine toxicology results available.
Measure: Count of Participants; unit: Participants
Arm/Group | Integrated Care Van (ICV) | Control
Number analyzed (Participants) | 267 | 242
Participants
  Have a negative urine drug test for selected drugs | 42 | 25
  Have a positive urine drug test for selected drugs | 225 | 217

12. Secondary Outcome: Sharing Injection Equipment
Description: This outcome will be assessed in all participants at all time points. The score is based on self-report and ranges from 0 to 2 with higher scores indicating riskier behavior.
  Participants who did not share needle/syringe or cotton/cooker in the prior 6 months are counted and assigned a score=0; those who shared cotton/cooker but did not share needle/syringes in the prior 6 months are counted and assigned a score=1; those who shared needle/syringes in the prior 6 months are counted and assigned a score=2. The counts of participants will be reported for this outcome measure and the associated score will be factored into the primary composite outcome.
Time Frame: Between 6 months prior to and the V7 follow-up visit at 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Integrated Care Van (ICV) | Control
Number analyzed (Participants) | 268 | 243
Participants
  Did not share needle/syringe or cotton/cooker in the prior 6 months | 202 | 175
  Shared cotton/cooker but did not share needle/syringes in the prior 6 months | 21 | 23
  Shared needle/syringes in the prior 6 months | 45 | 45

13. Secondary Outcome: Non-fatal Overdose
Description: This outcome will be assessed in all participants at all time points. The score is based on self-report, and ranges from 0 to 1 with higher scores indicating adverse outcome.
  Participants who do not report a non-fatal drug overdose in the prior 6 months are counted and assigned a score=0; those who report a non-fatal drug overdose in the prior 6 months are counted and assigned a score=1. The counts of participants will be reported for this outcome measure and the associated score will be factored into the primary composite outcome.
Time Frame: Between 6 months prior to and the V7 follow-up visit at 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Integrated Care Van (ICV) | Control
Number analyzed (Participants) | 268 | 243
Participants
  Do not report a non-fatal drug overdose in the prior 6 months | 230 | 210
  Report a non-fatal drug overdose in the prior 6 months | 38 | 33

14. Secondary Outcome: Emergency Department (ED) Use
Description: This outcome will be assessed in all participants at all time points. The score is based on self-report, and ranges from 0 to 1, with higher scores indicating adverse outcome.
  Participants with no ED visits in the prior 6 months are counted and assigned a score=0; those with 1 or more ED visits in prior 6 months are counted and assigned a score=1. The counts of participants will be reported for this outcome measure and the associated score will be factored into the primary composite outcome.
Time Frame: Between 6 months prior to and the V7 follow-up visit at 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Integrated Care Van (ICV) | Control
Number analyzed (Participants) | 268 | 243
Participants
  No ED visits in the prior 6 months | 166 | 144
  With 1 or more ED visits in prior 6 months | 102 | 99

15. Secondary Outcome: HIV Seroconversion
Description: This outcome will be assessed in participants who were HIV-negative at baseline, at follow-up time points. The score is based biomarker testing, and ranges from 0 to 1 with higher scores indicating adverse outcome.
  Participants who remain HIV seronegative at follow-up visits are counted and assigned a score=0; those who seroconvert for HIV are counted and assigned a score=1. The counts of participants will be reported for this outcome measure and the associated score will be factored into the primary composite outcome.
Time Frame: Between baseline visit and the V7 follow-up visit at 7 months
Population: Subset of participants who were HIV-negative at baseline and completed the V7 follow-up visit
Measure: Count of Participants; unit: Participants
Arm/Group | Integrated Care Van (ICV) | Control
Number analyzed (Participants) | 237 | 211
Participants
  HIV seronegative at follow-up visits | 236 | 210
  Seroconvert for HIV | 1 | 1

16. Secondary Outcome: HCV Seroconversion
Description: This outcome will be assessed in participants who were HCV seronegative at baseline, at follow-up time points. The score is based biomarker testing, and ranges from 0 to 1 with higher scores indicating adverse outcome.
  Participants who remain HCV seronegative at follow-up visits are counted and assigned a score=0, those who seroconvert for HCV are counted and assigned a score=1. The counts of participants will be reported for this outcome measure and the associated score will be factored into the primary composite outcome.
Time Frame: Between baseline visit and the V7 follow-up visit at 7 months
Population: Subset of population who were HCV-negative at baseline and completed a V7 follow-up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Integrated Care Van (ICV) | Control
Number analyzed (Participants) | 88 | 111
Participants
  HCV seronegative at follow-up visits | 87 | 105
  Seroconvert for HCV | 1 | 6

17. Secondary Outcome: Mortality Rate
Description: This outcome will be assessed in all participants at all follow-up time points. The score is based on medical record review or National Death Index, and ranges from 0 to 1 with higher scores indicating adverse outcome.
  Participants who are alive are counted and assigned a score=0, those who have died are counted and assigned a score=1. The counts of participants will be reported for this outcome measure and the associated score will be factored into the primary composite outcome.
Time Frame: Between baseline visit and the V7 follow-up visit at 7 months
Population: Subset of participants who completed the V7 follow-up visit and participants who died prior to completing the V7 follow-up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Integrated Care Van (ICV) | Control
Number analyzed (Participants) | 272 | 250
Participants
  Alive | 268 | 243
  Died | 4 | 7

18. Other Pre Specified Outcome: Participants Who Completed Qualitative Assessments
Description: To provide context and identify facilitators and barriers to the intervention, investigators will conduct qualitative assessments. First, investigators will conduct in-depth interviews (IDIs) with ~ 30 PWID participants. The interview will explore accessibility, coverage, and barriers accessing the services in question. Second, investigators will conduct IDIs with Baltimore City Health Department (BCHD) staff who work on either the existing SSP van or the newly created ICV (N~12). The interview will explore feasibility, perceived benefits and challenges of offering services in the field, and changes in perceptions after intervention roll-out on the ICV. Third, conduct IDIs with BCHD and Maryland Department of Health and Mental Hygiene (DHMH) officials and managers who are involved in PWID services (N~10). The interview will explore feasibility, and perceived benefits and challenges of offering services in the field on the ICV. Investigators will digitally record the interviews.
Time Frame: 12 months
Population: Participants who completed qualitative in-depth interviews
Measure: Count of Participants; unit: Participants
Groups:
- Stakeholders: This group was comprised of community, program, and health department stakeholders including care van staff, needle exchange service staff, and city and state health department officials.
- Care Van Clients: This group was comprised of clients who received services from the integrated care van intervention.
- Non-clients: This is a group of individuals who would have been eligible to receive services from the integrated care van intervention but had not engaged in care at that mobile service clinic.
Arm/Group | Stakeholders | Care Van Clients | Non-clients
Number analyzed (Participants) | 18 | 16 | 15
Participants | 18 | 16 | 15

19. Other Pre Specified Outcome: Costs and Cost Effectiveness
Description: In accordance with the recommendations of the 2nd US Panel on Cost-Effectiveness in Heath and Medicine, we will: inventory and value the resources consumed in the ICV intervention; estimate intervention effectiveness in regards to viral suppression, HIV infections averted, HCV treatment, and MAT use; estimate treatment costs averted and Quality-adjusted life years saved for each type of effectiveness; and determine whether the ICV is cost-saving, cost-effective, or not cost-effective.
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Each participant was followed for adverse event data during study visits. Death data was collected for all participants through the end of the Pre-COVID V14 Follow-up window for participants followed from the first 4 sites and through the end of the Post-COVID V14 Follow-up window for participants in the last 8 sites (maximum of 4 years).
Description: These research procedures are minimal risk (involve only a blood draw), do not include a drug or medical device, and the intervention was being rolled out by the BCHD. Finally, the study population (active PWID) have relatively high rates of mortality and morbidity compared to the general public. Given these considerations, our reporting obligations for the trial focus only on events that are more likely than not to be associated with study procedures (study visits or key-informant interviews).
Arm/Group | Integrated Care Van (ICV) | Control
All-Cause Mortality (participants affected / at risk) | 24/360 | 31/360
Serious Adverse Events (participants affected / at risk) | 24/360 | 31/360
Other Adverse Events (participants affected / at risk) | 0/360 | 0/360
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Integrated Care Van (ICV) (N=360) | Control (N=360)
Death (General disorders) | 24 (24) | 31 (31)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/74/NCT03567174/Prot_SAP_000.pdf